CLINICAL TRIAL: NCT03282695
Title: Ozone Therapy in Patients on Waiting List for Surgery Due to Disc Herniation: Prospective, Post-authorization Study
Acronym: O3HDCIRUGIA
Status: Active, not recruiting | Type: Observational
Sponsor: Bernardino Clavo, MD, PhD (Other)
Collaborators: Servicio Canario de Salud (Other); Red de Investigación en Servicios de Salud en Enfermedades Crónicas (Other); Instituto de Salud Carlos III (Other Government); Colegio Oficial de Médicos de Las Palmas (Unknown)
Responsible Party: Sponsor-Investigator, Bernardino Clavo, MD, PhD, MD. PhD, Dr. Negrin University Hospital
Organization: Dr. Negrin University Hospital (Other)
Other Study IDs: BCV-OZO-2016-01
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Lumbar Herniated Disc
Keywords: Disc Herniation; Lumbar Herniated Disc; Ozone Therapy
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Surgery: Patients on waiting list for surgery (by discectomy/microdiscectomy) who reject ozone infiltration during waiting time.
  These patients will receive standard pain treatment until the planned surgery.
- Ozone: Patients on waiting list for surgery (by discectomy/microdiscectomy) who accept treatment by ozone infiltration during waiting time.
  These patients will be treated primarily by ozone therapy: Infiltration of intradiscal O3/O2 + foraminal infiltration of O3/O2 + corticoid + anesthetic.
  These patients will receive standard pain treatment until the planned surgery.

SUMMARY:
The main objective of this study is to estimate the cost-effectiveness of ozone therapy in patients on the waiting list for surgery due to disc herniation.

DETAILED DESCRIPTION:
A cohort study (patients on the waiting list for surgery due to herniated disc) will be carried out, to which the treatment with ozone will be offered, without giving up the planned surgical intervention.

The main objective of this prospective, post-authorization follow-up study is to estimate the cost-effectiveness of ozone therapy (compared to standard care) in patients with disc herniation waiting for surgery (by microdiscectomy). Besides utilities of patients with disc herniation on a waiting list for surgery will be estimated, social/economic burden of disc herniation will be quantified and a decision aid will be developed and applied.

The main outcome measures are "Direct hospital cost", "Percentage of executed surgeries" and "Change in sciatic pain". In addition, data on health-related quality of life and resource utilization will be collected which will permit to estimate the incremental cost-effectiveness ratio (ICER), comparing incremental costs and quality adjusted life years (QALY).

The variables will be collected at the beginning, on the day of treatment and at 1, 3, 6, 12 and 24 months. The enrollment period will be 24 months. The follow-up period will be 24 months.

The results of the study will allow a better understanding of the value of ozone therapy in the management of patients on the waiting list for herniated disc surgery. In addition, it will contribute to the development of a more patient-centered health system.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a herniated and not calcified lumbar disc that presents as: not migrated protrusion and/or extrusion.
* Evaluated and diagnosed by the Neurosurgery Department, having been chosen as an appropriate candidate for surgery consisting in discectomy or microdiscectomy, after meeting the following two criteria: 1) Sciatic pain, with a visual analogue scale (VAS) intensity ≥ 5, despite 6 weeks of conservative management, wether it exists lumbar pain or not and 2) Radiating pain that matches the MRI image showing one or more herniated discs (not to be considered those patients with two herniated discs and symptoms attributable to only one of the herniated discs).
* Included in the surgery waiting list for a discectomy or microdiscectomy.
* Patients who have signed and dated the study 's specific informed consent.

Exclusion Criteria:

* Patients who do not meet all the inclusion criteria.
* Calcified and/or migrated herniated disc, and/or with a severe neurological deficits (cauda equine syndrome).
* Herniated disc with surgical indication of laminectomy and/or arthrodesis (massive extrusion, sign of instability or other conditions under the neurosurgeon judgment).
* Relevant clinical paresis that does not improve despite 6 weeks of full conservative management (patients with severe pain and mild paresis that only shows up in the physical exam are not to be excluded, but those who present with paresis as the main symptom -"clinically relevant"- must be).
* Simultaneous symptomatic cervical or dorsal herniated discs.
* Previous lumbar spine surgery.
* Concomitant spine conditions that may be causing symptoms or have indication for surgery (such as fractures or tumors).
* Known allergy to ozone.
* Those who are uncapable to fill in the scales used to measure variables in the study, like the visual analogue scale (VAS), Roland-Morris and SF-12 questionnaires.
* Those who are unable or do not wish to fulfill the study 's protocol (answer questions to collect the data).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with symptomatic lumbar herniated disc in whom conservative medical management has failed and: 1) in whom discectomy or microdiscectomy is indicated, 2) have been included in surgery waiting list by the Neurosurgery Department, 3) who meet criteria for potential benefit with ozone therapy and 4) who accept participating in the study by answering/filling in the specific study questionnaires (wether they accept or not the ozone therapy).
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Direct Hospital Cost for patients included on waiting list for surgery due to disc herniation. | 24 months
  Euros
Percentage of surgeries finally performed. | 24 months
  Percentage of surgeries performed after enrollment
Change from Baseline in sciatic pain at 12 months | 12 months
  Visual Analogic Scale (VAS)
Change from Baseline in sciatic pain at 24 months | 24 months
  Visual Analogic Scale (VAS)

SECONDARY OUTCOMES:
Change from Baseline in sciatic pain at 6 months | 6 months
  Visual Analogic Scale (VAS)
Change from Baseline in lumbar pain at 6 months | 6 months
  Visual Analogic Scale (VAS)
Change from Baseline in lumbar pain at 12 months | 12 months
  Visual Analogic Scale (VAS)
Change from Baseline in lumbar pain at 24 months | 24 months
  Visual Analogic Scale (VAS)
Number of hospital stay days | 24 months
  Number of hospital stay days
Restriction of everyday activities | 24 months
  Spanish version of Roland-Morris questionnaire
Quality of life by 12-Item Short Form Survey (SF-12) | 24 months
  SF-12 questionnaire
Quality of life by the five-level version of the EuroQol five-dimensional (EQ-5D-5L) questionnaire | 24 months
  EQ-5D-5L questionnaire
Loss of labour productivity | 24 months
  Off work days (if applicable)
Time to resume normal activity | 24 months
  Days
Direct sanitary and non-sanitary costs incurred out of hospital. | 24 months
  Euros
Adverse effects | 24 months
  Number of serious adverse effects
Time from inclusion on waiting list for surgery to completion of the procedure. | 24 months
  Days

CONTACTS AND LOCATIONS:
Overall Officials: Bernardino Clavo, MD, PhD, Study Chair — Dr. Negrín University Hospital, Las Palmas, Spain; Pedro G. Serrano-Aguilar, MD, PhD, Study Director — Servicio de Evaluación. Servicio Canario de Salud. Spain; Renata Linertová, MD, PhD, Principal Investigator — Fundación Canaria de Investigación Sanitaria (FUNCANIS); Adam Szolna, MD, PhD, Principal Investigator — Dr. Negrín University Hospital, Las Palmas. Spain
Locations (1):
- Dr. Negrin University Hospital, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hansson E, Hansson T. The cost-utility of lumbar disc herniation surgery. Eur Spine J. 2007 Mar;16(3):329-37. doi: 10.1007/s00586-006-0131-y. Epub 2006 May 9. PMID 16683121
- [Background] Luhmann D, Burkhardt-Hammer T, Borowski C, Raspe H. Minimally invasive surgical procedures for the treatment of lumbar disc herniation. GMS Health Technol Assess. 2005 Nov 15;1:Doc07. PMID 21289928
- [Background] Magalhaes FN, Dotta L, Sasse A, Teixera MJ, Fonoff ET. Ozone therapy as a treatment for low back pain secondary to herniated disc: a systematic review and meta-analysis of randomized controlled trials. Pain Physician. 2012 Mar-Apr;15(2):E115-29. PMID 22430658
- [Background] Sherman J, Cauthen J, Schoenberg D, Burns M, Reaven NL, Griffith SL. Economic impact of improving outcomes of lumbar discectomy. Spine J. 2010 Feb;10(2):108-16. doi: 10.1016/j.spinee.2009.08.453. Epub 2009 Oct 12. PMID 19819761
- [Background] Tosteson AN, Skinner JS, Tosteson TD, Lurie JD, Andersson GB, Berven S, Grove MR, Hanscom B, Blood EA, Weinstein JN. The cost effectiveness of surgical versus nonoperative treatment for lumbar disc herniation over two years: evidence from the Spine Patient Outcomes Research Trial (SPORT). Spine (Phila Pa 1976). 2008 Sep 1;33(19):2108-15. doi: 10.1097/brs.0b013e318182e390. PMID 18777603
- See also: Report (June 2016) about Ozone therapy in disc herniation, from the Health Technology Assessment (HTA) Unit, Canary Health Service, Spain — http://www3.gobiernodecanarias.org/sanidad/scs/content/4c7be1f8-a10e-11e6-a33b-757951c5b2fa/Informe_Ozonoterapia_SESCS%202016.pdf